CLINICAL TRIAL: NCT01647503
Title: Identification of Differentially Expressed Proteins in Parathyroid Tumors and Their Clinical Correlation With the Disease
Brief Title: Differentially Expressed Proteins in Sporadic Parathyroid Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Sanjay K. Bhadada, Associate Professor, Dept of Endocrinology, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Other Study IDs: parathyroid tumorigenesis
Record Dates: First submitted 2012-07-18; First posted 2012-07-23 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Primary Hyperparathyroidism; Hypercalcemia
Keywords: parathyroid gland; primary hyperparathyroidism; proteins
MeSH Terms: conditions — Hyperparathyroidism, Primary; Hypercalcemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Tumor group: Parathyroid adenoma, hyperplasia and carcinoma
- Normal: Normal parathyroid samples

SUMMARY:
Primary hyperparathyroidism (PHPT) is one of the common endocrine disorders. The major clinical symptoms involve stones, bones, abdominal groans and psychiatric moans. Increased parathyroid cell proliferation and decreased calcium-mediated control of the PTH secretion are characteristic findings. The most common cause of PHPT is adenoma followed by hyperplasia and carcinoma.The molecular mechanisms involved in parathyroid tumorigenesis are partially known. Few genes have been identified and their roles are under study.

The genes which are under study by different groups are unable to give a definite direction towards the understanding of parathyroid tumorigenesis and the mechanism involved in overgrowth of parathyroid tissue. So identifying different proteins and their regulation pattern from adenomas to carcinomas will be the initial steps towards understanding the proteins involved in tumorigenesis of parathyroid tissues. By using proteomics approach one can generate protein level information. In this study, using a combined approach based on 2 D gel electrophoresis and mass spectrometry (MS), the investigators propose to study a comparative proteomics to examine the changes of protein profiles in parathyroid tumor tissues with normal and hyperplasic parathyroid tissues. This work plan will help us to understand differentially expressed proteins in patients with PHPT. This will help in understanding the disease and identifying better diagnostic and curative measures of the disease. The investigators are also planning to access nuclear morphometry changes in sporadic parathyroid tumors. It will help in establishing cellular and nuclear change pattern variations from normal to parathyroid tumors.

DETAILED DESCRIPTION:
Subjects:

All the PHPT patients attending outdoor patient clinic of Endocrinology and General Surgery department of Nehru Hospital, PGIMER, Chandigarh will be enrolled in this study.

Sample collection:

A parathyroid tissue sample will be taken from the patients undergoing for parathyroidectomy. Samples will be collected immediately after surgery, snap frozen and stored at -80oC until use. In addition 10 ml of blood will also be taken from these patients for estimating biochemical parameters.

Controls:

Normal parathyroid gland will be used as control and it will be obtained from patient undergoing thyroidectomy for multinodular goiter as an elective procedure at the institute.

ELIGIBILITY:
Inclusion Criteria:

* PHPT patients with parathyroid adenoma, hyperplasia and carcinoma

Exclusion Criteria:

* Patients with family history, HPT-JT syndrome and familial isolated hyperparathyroidism

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients visiting the hospital for hypercalcemia, bone pain, renal problems and other symptoms related to primary hyperparathyroidim will be consider. Investigations and clinical symptoms will be confirmed for primary hyperpathyroidism. Finally if patient suggested for surgery then he will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Differentially expressed proteins in parathyroid adenomas tissue samples | At the end of three years of the study

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Kr Bhadada, DM, Principal Investigator — Associate Professor, Department of Endocrinology, PGIMER Chandigarh India
Locations (1):
- PGIMER, Chandigarh, Uttarakhand, India